CLINICAL TRIAL: NCT05156359
Title: Idiopathic Scoliosis and Orthodontic Treatment
Acronym: SITO
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8049
Record Dates: First submitted 2021-10-13; First posted 2021-12-14 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Scoliosis
Keywords: Idiopathic scoliosis; Orthodontic Treatment; spinal dysmorphism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scoliotic pathology remains to this day little known, on the one hand in its etiologies but also in its various implications and possible associations. One of the notable questions found in the literature is concerned with the link between idiopathic scoliosis and the stomatognathic system. This question arises from the study of the anatomy and function of its two entities.

The aim of the study is to determine the frequency of orthodontic treatment in adolescents with idiopathic scoliosis, and to compare it with that of adolescents without spinal dysmorphism.

ELIGIBILITY:
Inclusion criteria:

* Adult and child (age ≥ 12 years)
* Be carriers of idiopathic scoliosis confirmed by X-ray.
* Have reached bone maturity (Risser 4 and more)
* Adult who has not expressed, after information, the reuse of his data for the purposes of this research
* - Child and Holders of parental authority who have not expressed, after information, the reuse of their data for the purposes of this research

Exclusion criteria:

* Refusal to participate in the study
* Association with another orthopedic pathology
* Adult patients under guardianship or crater or under the protection of justice

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children (age ≥ 12 years) with idiopathic scoliosis confirmed by X-ray.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Determination of the frequency of wearing orthodontic treatment in idiopathic scoliosis adolescents, and compare it with that of adolescents without spinal dysmorphism. | Files analysed retrospectively from January 01, 2020 to August 31, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie Orthopédique Pédiatrique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France